CLINICAL TRIAL: NCT05696938
Title: Improved Skin Whitening Outcomes Associated With Nicotinamide Fortified Consumption in 30 to 50-Year-old Women, a Double Blind, Control and Randomized Study
Brief Title: Improved Skin Whitening Outcomes Associated With Nicotinamide Fortified Consumption in 30 to 50- Year-old Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Precision Health Food Technology Co. Ltd., (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-SM-11-WL-001
Record Dates: First submitted 2022-12-27; First posted 2023-01-25 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Skin Darken
Keywords: skin whitening; nicotinamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Wonderlab Nicotinamide Drink (Active Comparator): 25ml/bottle, containing the following ingredients per 25ml serving:
  * Nicotinamide 0.39 mg
  * Vitamins C 300 mg
  * Hyaluronic acid 50 mg
  * Tomato powder 120 mg
  Interventions: Dietary Supplement: Wonderlab Nicotinamide Drink
- Ordinary Drink (Placebo Comparator): 25ml/bottle, containing the following ingredients per 25ml serving:
  * Litchi juice 0.7 g
  * Erythritol 2 g
  * Pectin 0.25 g
  Interventions: Dietary Supplement: Ordinary Drink

INTERVENTIONS:
Dietary Supplement: Wonderlab Nicotinamide Drink — Participants in this arm will use a bottle of 25ml each time, twice a day, for 2 months.
  Arms: Wonderlab Nicotinamide Drink
Dietary Supplement: Ordinary Drink — Participants in this arm will use a bottle of 25ml each time, twice a day, for 2 months.
  Arms: Ordinary Drink

SUMMARY:
The goal of this clinical trial is to study whether the products with nicotinamide fortified could improve skin whitening in 30 to 50-year-old women.

Partipants will be randomly assigned to two study groups and use products (study product plus nicotinamide supplement and placebo product without nicotinamide supplement) for 2 months, twice a day.

Researchers will compare the two groups whether there are significant improvement in skin whitening via skin measurement and analysis systems.

DETAILED DESCRIPTION:
This study is two arms, randomized, double-blind controlled trial. 70 eligible partipants at two study sites will be enrolled and use randomly assigned products (study product plus nicotinamide supplement and placebo product) for 2 months. Participants will visit the study site for three times on baseline day, day 30, and day 60, all relevant data will be captured, measured via professional skin equipment system and recorded in the data management system. At the end of study, the explantory and statisitcal analysis will be conducted to validate the assumption that the using products with nicotinamide fortified could improve skin whitening in 30 to 50-year-old women.

ELIGIBILITY:
Inclusion Criteria:

* Chinese females, age between 30-50;
* Be in general good health;
* Understand the test procedure, read, and sign an appropriate Informed Consent Form indicating their willingness to participate;
* Be free from tattoos, cuts, scratches, abrasions, scars, uneven skin tone, sunburn, excessive tanning, open wounds, excessive hair, and visible skin disease on the inner forearm;
* Has the skin lightness parameter L* < 60 on the inner forearm the beginning of the product application phase;
* Willing and able to follow all study directions, undergo skin examination and commit to all follow-up visits;
* Individuals in good general health (no physical required) and not taking any prescribed medicines (except for oral contraceptives or asthma inhalers) that could interfere with the conduct of the study;
* Agree to not use any other creams, lotions, moisturizers on the face, other than what is provided for the duration of the study;
* Agree to refrain from wearing make-up (such as foundation, eye shadow, lipstick etc.) or any skin care products on the face on the study visits;
* Agree to avoid washing the treatment site area for two hours following product application and agree to avoid washing appliances (i.e., sponge, wash cloth, loofah, etc.).

Exclusion Criteria:

* Have used any skin lightening /anti-aging benefits products at least one month before this study
* Subject having done facial injections and/or aesthetic surgery.
* Be involved in any aspect of test administration, i.e., evaluating or overseeing activities related to product.
* Have participated in any clinical study involving the test sites within the previous 6 months, or is subject participating in any clinical study concurrently.
* Have a history of any type of bottlecer, including but not limited to any type of skin bottlecer (squamous or basal cell carcinoma at the treatment site) or history of malignant melanoma at any body site.
* Have a history of skin disease or the presence of a skin condition on the test sites that the Investigator feels would interfere with the study.
* Be taking antihistamines (> 3x/week) or anti-inflammatory (> 8x/week) on a regular basis, or has the subject taken systemic or topical steroidal medications within 4 weeks of study enrolment.
* Have any of the following conditions or factors that the investigator believes may affect the response of the skin or the interpretation of the test results, including, but not limited to, diabetes, pregnancy, lactation.
* Have any cuts/abrasions on the test site at baseline.
* Have had a suspicious skin lesion removed by a dermatologist at any time.
* The subject is an employee of sponsor or the site conducting the study.

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — must be momen of 30 to 50 years old
Enrollment: 70 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
Skin Brightness | baseline day 0, day 30, day 60
  The changes of the skin brightness by Spectrophotometer CM2600D

SECONDARY OUTCOMES:
Skin Barrier | baseline day 0, day 30, day 60
  The changes of skin barrier in terms of TEWL (Trans Epidermal Water Loss) via Aquaflux F200
Skin Hydration | baseline day 0, day 30, day 60
  The changes of skin hydration by Corneometer CM 825
Skin Gloss | baseline day 0, day 30, day 60
  The changes of skin gloss by Glossmeter
Skin Radiance Scale | baseline day 0, day 30, day 60
  The changes of skin radiance scale (0-9) assessed in three aspects (Radiant Lumimous,Shallowness, and Dullness) by professionals

CONTACTS AND LOCATIONS:
Overall Officials: Yun Wang, MD, Principal Investigator — NO. 9 Hospital affiliated to Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Ai'er Hospital, Shanghai, Shanghai Municipality
  - SPRIM Central Lab, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bains P, Kaur M, Kaur J, Sharma S. Nicotinamide: Mechanism of action and indications in dermatology. Indian J Dermatol Venereol Leprol. 2018;84(2):234-237. doi: 10.4103/ijdvl.IJDVL_286_17. No abstract available. PMID 29405129
- [Background] Zhao J, Liu Z, Zhang C, Wu J, Huang N, Du Y, Xiang L. Dynamic evaluation of an in vivo postinflammatory hyperpigmentation model using reflectance confocal microscopy and spectrophotometry. J Cosmet Dermatol. 2021 Sep;20(9):2950-2962. doi: 10.1111/jocd.13932. Epub 2021 Feb 13. PMID 33394548
- [Background] Shariff R, Du Y, Dutta M, Kumar S 5th, Thimmaiah S, Doraiswamy C, Kumari A, Kale V, Nair N, Zhang S, Joshi M, Santhanam U, Qiang Q, Damodaran A. Superior even skin tone and anti-ageing benefit of a combination of 4-hexylresorcinol and niacinamide. Int J Cosmet Sci. 2022 Feb;44(1):103-117. doi: 10.1111/ics.12759. Epub 2022 Feb 1. PMID 34958693
- [Background] Wang L, Xu YN, Chu CC, Jing Z, Chen Y, Zhang J, Pu M, Mi T, Du Y, Liang Z, Doraiswamy C, Zeng T, Wu J, Chen L. Facial Skin Microbiota-Mediated Host Response to Pollution Stress Revealed by Microbiome Networks of Individual. mSystems. 2021 Aug 31;6(4):e0031921. doi: 10.1128/mSystems.00319-21. Epub 2021 Jul 27. PMID 34313461
- [Background] Du Y, Doraiswamy C, Mao J, Zhang Q, Liang Y, Du Z, Vasantharaghavan R, Joshi MK. Facial skin characteristics and concerns in Indonesia: A cross-sectional observational study. Skin Res Technol. 2022 Sep;28(5):719-728. doi: 10.1111/srt.13189. Epub 2022 Jul 4. PMID 35785442